CLINICAL TRIAL: NCT01331915
Title: Phase I/II Study of Therapeutic Vaccination With Escalating Doses of Theravac®, a Proteinic Vector Targeting Dendritic Cells Coupled to a Melanoma Antigen, in Patients With Advanced Metastatic Melanoma.
Brief Title: Safety and Toxicity Study of Vaccination for Advanced Metastatic Melanoma Patients
Acronym: THERAVAC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUC 09-003; 2009-014651-77 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-04-08 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma; Safety; Theravac vaccine; HLA-A2 typing; Tyrosinase.A2 gene expression
MeSH Terms: conditions — Melanoma

ARMS (1):
- Theravac (Experimental): Theravac® is a recombinant adenylate cyclase toxin from Bordetella pertussis that has been detoxified by mutation of its catalytic domain, and which has been coupled to the Tyrosinase.A2 epitope YMDGTMSQV.
  Interventions: Biological: Theravac

INTERVENTIONS:
Biological: Theravac — Three groups with three doses (50 - 150 - 250 mcg), four times every three weeks.
  Injection: intradermally and subcutaneously.

SUMMARY:
In this phase I study, the investigators want to vaccine with THERAVAC® (an inactivated toxin coupled to melanoma antigen) some patients with advanced metastatic melanoma disease.

The primary objective is to analyze the safety of the inreasing doses of vaccine.

The secondary objective is to document whether this vaccine can induce tumor regression in immunized patients.

DETAILED DESCRIPTION:
There are three treatment cohorts and the inclusion of patients in governed by the dose-limiting toxicities in the previous cohort.

* the first three patients will receive a dose of 50 µg of Theravac®
* second cohort of three patients will receive a dose of 150 µg Theravac®
* the third cohort of three patients will receive a dose of 250 µg Theravac® and eventually a total of 14 patients will complete the step with the highest dose.

All the patients will receive four immunizations every three weeks in two intradermal sites and in two subcutaneous sites.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven cutaneous, uveal or mucosal melanoma.
2. Melanoma must be metastatic. The origin of the primary could be cutaneous, uveal or mucosal and any metastatic stage is accepted, except if brain or leptomeningeal localizations are present, or if plasma LDH are elevated more than 1.5 normal upper values (see also below).
3. HLA-A2 positive.
4. The melanoma must express the tyrosinase gene (positive RT-PCR on a frozen pre-immune tumor sample) (see Appendix B).
5. At least one measurable or non-measurable tumor lesion (see Section 8.1).
6. Expected survival of at least 3 months.
7. Karnofsky performance scale ≥70 or WHO performance status of 0 or 1 (see Appendix C).
8. Vital laboratory parameters should be within normal range, except for the following laboratory parameters, which must be within the ranges specified:

   Lab Parameter Range Hemoglobin ≥ 10 g/dl or ≥ 6,25 mmol/l Granulocytes ≥ 1,500/µl Lymphocytes ≥ 700/µl Platelets ≥ 100,000/µl Serum creatinin ≤ 2.0 mg/dl or ≤ 177 μmol/l Serum bilirubin ≤ 2.0 mg/dl or ≤ 34.2 μmol/l ASAT and ALAT ≤ 2 x the normal upper limits LDH ≤ 1.5 x the normal upper limit.
9. Viral serology:

   * HIV (human immunodeficiency virus): negative antibodies.
   * HBV (hepatitis B virus): negative antigens; antibodies may be positive.
   * HCV (hepatitis C virus): negative antibodies.
10. Age ≥ 18 years
11. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Previous treatment with more than one regimen of systemic chemotherapy, combined or not with non-specific immunotherapy such as interferon alpha or interleukins. Chemoimmunotherapy or radiotherapy must be stopped within the preceding 4 weeks (6 weeks for nitrosoureas and mitomycin C).
2. Previous treatment with a vaccine known or likely to contain the Tyrosinase.A2 epitope YMDGTMSQV.
3. Clinically significant heart disease (NYHA Class III or IV) i.e. NYHA class 3 congestive heart failure; myocardial infarction within the past six months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias.
4. Active immunodeficiency or autoimmune disease. Vitiligo is not an exclusion criterion.
5. Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders, or other conditions requiring concurrent medications not allowed during this study.
6. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
7. Allergy to kanamycin (used in the preparation of the recombinant protein) or to any other aminoglycoside antibiotic.
8. Lack of availability for immunological and clinical follow-up assessments.
9. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
10. Pregnancy or breastfeeding.
11. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
To analyze the safety and toxicity of increasing doses of Theravac® in patients with advanced metastatic melanoma | the first 3 months of treatment
  The toxicity will be assess after the treatment (3 months) for the first three patients of each group.
To determine whether these immunizations result in a detectable immune response | Up to 24 weeks
  PBMC will be obtained from the buffy-coat of 500 ml of venous blood or from 100 ml of venous blood collected before and after immunization.

SECONDARY OUTCOMES:
To document whether this vaccine can induce tumor regression in immunized patients. | at week 12
  The NEW RECIST criteria when applicable. For patients with only non-measurable lesion(s) at study entry, tumor response will be assessed descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Baurain, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc, Centre du Cancer
Locations (1):
- Cliniques universitaires Saint-Luc, Centre du Cancer, Brussels, Brussels Capital, Belgium